CLINICAL TRIAL: NCT04586348
Title: Prenatal Iodine Supplementation and Early Childhood Neurodevelopment
Acronym: PoppiE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: South Australian Health and Medical Research Institute (Other)
Collaborators: Women's and Children's Hospital, Australia (Other Government); Flinders Medical Centre (Other Government); Mater Mothers' Hospital (Other); The Royal Women's Hospital (Unknown); Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Karen Best, Senior Research Fellow, South Australian Health and Medical Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PoppiE
Record Dates: First submitted 2020-09-30; First posted 2020-10-14 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy Related; Neurodevelopmental Disorders; Nutrition Disorder, Fetal
Keywords: Iodine; Supplementation
MeSH Terms: conditions — Neurodevelopmental Disorders; Fetal Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: A multi-centre, randomised, controlled, clinician, researcher and participant blinded trial with two parallel groups. An independent statistician not otherwise involved in the study or data analysis will generate and keep the randomisation schedule. The computer-generated schedule will allocate women to intervention or control groups in the ratio of 1:1 using randomly permuted blocks of size 6 and 8, with stratification for state of enrolment.
  Randomisations will be performed by approved study staff via a secure web-based randomisation service.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Intervention and Control supplements will be packaged by Factors Group of Companies and labelled by contracted pharmaceutical personnel who are not involved in the trial. Study supplement bottles will be identified only by the blinded Product ID to match the randomisation schedule prepared by an independent statistician.
  Research Personnel will access the Randomisation Module in REDCap and women will be allocated a random, unique, re-identifiable randomisation ID. Women will be issued with supplements labelled to match their unique assigned code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Iodine Supplement (Experimental): Iodine (potassium iodide) 20 μg Beta carotene (All trans-beta- carotene) 1500 μg; Vitamin E (dl-alphatocopheryl acetate) 13.5 mg AT; Vitamin D3 (cholecalciferol) 10 μg; Vitamin C (ascorbic acid granular) 60 mg; Niacinamide 18 mg; Pantothenic acid (calcium d- pantothenate) 6 mg; Vitamin B6 (DC pyridoxine hydrochloride) 1.9 mg; Vitamin B1 (thiamine mononitrate) 1.4 mg; Vitamin B2 (riboflavin) 1.4 mg; Biotin 30 μg; Vitamin B12 (methyl-cobalamin) 2.6 μg; Folic Acid 0.4 mg; Levomefolic acid 0.1 mg; Calcium (carbonate DC) 250 mg; Magnesium (oxide granular) 50 mg; Iron (ferrous fumarate) 20 mg; Zinc (oxide) 10 mg; Manganese (sulphate) 2 mg; Copper (sulphate) 1 mg; Selenium (rice chelate) 30 μg
  Interventions: Combination Product: Low Iodine Supplement
- Standard Iodine Supplement (Active Comparator): Iodine (potassium iodide) 200 μg Beta carotene (All trans-beta- carotene) 1500 μg; Vitamin E (dl-alphatocopheryl acetate) 13.5 mg AT; Vitamin D3 (cholecalciferol) 10 μg; Vitamin C (ascorbic acid granular) 60 mg; Niacinamide 18 mg; Pantothenic acid (calcium d- pantothenate) 6 mg; Vitamin B6 (DC pyridoxine hydrochloride) 1.9 mg; Vitamin B1 (thiamine mononitrate) 1.4 mg; Vitamin B2 (riboflavin) 1.4 mg; Biotin 30 μg; Vitamin B12 (methyl-cobalamin) 2.6 μg; Folic Acid 0.4 mg; Levomefolic acid 0.1 mg; Calcium (carbonate DC) 250 mg; Magnesium (oxide granular) 50 mg; Iron (ferrous fumarate) 20 mg; Zinc (oxide) 10 mg; Manganese (sulphate) 2 mg; Copper (sulphate) 1 mg; Selenium (rice chelate) 30 μg
  Interventions: Combination Product: Standard Iodine Supplement

INTERVENTIONS:
Combination Product: Low Iodine Supplement — Multivitamin and mineral supplement with reduced iodine
  Arms: Low Iodine Supplement
Combination Product: Standard Iodine Supplement — Multivitamin and mineral supplement with standard amount of iodine to match current leading brands of prenatal supplements
  Arms: Standard Iodine Supplement

SUMMARY:
A randomized controlled trial to determine the effect of reducing iodine from vitamin and mineral supplements for pregnant women who have adequate iodine intakes (>165 μg/d from food alone) on cognitive development of children at 24 months of age.

DETAILED DESCRIPTION:
It is known that severe iodine deficiency during pregnancy leads to profound intellectual disabilities in the child. Following results of a 2004 national survey of school-aged children showing that mild iodine deficiency had re-emerged in the south-eastern parts of Australia, the Australian government mandated the addition of iodine to salt used in bread making to increase population iodine intake. It is also recommended that all pregnant and lactating women take an additional iodine supplement containing 150 µg/d of iodine.

Since this time, further evidence has emerged from cohort studies that children born to women with high iodine intake (as well as low iodine intake) have poorer neurodevelopmental scores, suggesting that more tailored supplementation may be a better strategy. Our PoppiE trial will determine if limiting iodine supplementation in women who already consume adequate iodine from food, improves cognitive scores in early childhood.

A total of 754 pregnant women from around Australia who are ≤13 weeks of gestation will be enrolled and randomised to receive a standard prenatal vitamin and mineral supplement with a reduced amount of iodine (20 μg - intervention) or a standard prenatal vitamin and mineral supplement with 200 μg of iodine (control). The control supplement contains a level of iodine to match the amount in most commonly used vitamin and mineral supplements sold in Australia. Infant neurodevelopment at 24 months of age will be assessed using the Bayley-IV and conducted at participating centres or a location convenient to the family.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≤13 weeks of gestation.
* Consume greater than 165 µg/d of iodine from food alone based on our validated Iodine Specific Food Frequency Questionnaire (I-FFQ).
* English is main language spoken at home as child will need to understand and take instruction in English to participate in the neurodevelopmental assessment.
* Able to give informed consent.

Exclusion Criteria:

* Known history of thyroid disease.
* Previous child diagnosed with thyroid dysfunction.
* Carrying a fetus with a known or suspected congenital abnormality.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Infant Developmental quotient (DQ) | 24 months of age
  The Bayley Scales of Infant and Toddler Development, 4th Edition Cognitive Scale score has a mean of 100 and standard deviation of 15, where higher scores indicate a better outcome. As the Bayley scales are age-standardized scales the exact minimum and maximum score depends on the exact age of the child at the time of the assessment, hence we have instead provided the mean and standard deviation (as is the norm when reporting standardized psychometric assessments).

SECONDARY OUTCOMES:
Language development of infants using Bayley-IV | 24 months of age
  The Bayley Scales of Infant and Toddler Development, 4th Edition Language Scale score has a mean of 100 and standard deviation of 15, where higher scores indicate a better outcome.
Motor development of infants | 24 months of age
  The Bayley Scales of Infant and Toddler Development, 4th Edition Motor Scale score has a mean of 100 and standard deviation of 15, where higher scores indicate a better outcome.
Behavioral and emotional development | 24 months of age
  Behavioral and emotional development of infants using the Infant Toddler Social Emotional Assessment (ITSEA). The Infant-Toddler Social & Emotional Assessment scale has range of 0-100 where higher T scores indicate a worse outcome.
Health service utilization | 24 months of age
  Health service utilisation of children assessed through data linkage of the Medicare Benefits Schedule, Pharmaceutical Benefits Scheme to evaluate the cost effectiveness of the intervention.
Length of gestation | Birth
  The gestational age in days at birth (or other event of interest) will be determined from the estimated date of delivery using the equation [280 - (estimated date of delivery - date of birth)].
Infant Birth Anthropometrics | Birth
  Infant weight, length and head circumference will be analysed, using both the raw measurements and Z-scores for corresponding gestational age and sex, using means and standard deviations.
Admission to special care baby unit (level 2 nursery). | The neonatal period including birth to 28 days of age
  Any admission to a special care baby unit or level 2 nursery up to 28 days post birth.
Thyroid stimulating hormone (TSH) level | Within 5 days of birth
  Ascertained from Neonatal Screening Test
Infant Anthropometrics | 24 months of age
  Average weight, height and head circumference measurements at 24 months of age will be converted to z-scores using WHO growth standards. For preterm infants, corrected age at the time of the measurement rather than chronological age will be used in deriving the z-scores.

OTHER OUTCOMES:
Proportion of participants with pre-eclampsia | At any time throughout current pregnancy
  Clinical diagnosis of pre-eclampsia as recorded in the participants handheld record.
Proportion of participants with induction of labour and reason for induction. | Delivery
  As recorded in the participants handheld record.
Proportion of participants with postpartum hemorrhage | Within 24 hours of delivery of the infant
  Clinical diagnosis of postpartum hemorrhage as recorded in the participants handheld record.
Proportion of participants with gestational diabetes | At any time throughout current pregnancy
  Clinical diagnosis of gestational diabetes as recorded in the participants handheld record.
Proportion of participants with induced labour | Delivery
  As recorded in the participants handheld record.
Proportion of participants with vaginal delivery | Delivery
  Vaginal or caesarean delivery
Proportion of Maternal Adverse Events per group | From the date of randomization until delivery of the infant (up to 40 weeks)
  Side effects and tolerability of supplements will be assessed through routine data collection.
Proportion of Maternal Serious Adverse Events per group | From the date of randomization until the date of delivery (up to 40 weeks)
  Maternal admissions to intensive care during the intervention period. Maternal death in the intervention period.
Proportion of Fetal/Infant Serious Adverse Events | From the date of randomization until the infant is 24 months of age (up to 144 weeks)
  Fetal Mortality (after randomisation and prior to birth) including; miscarriage/terminations (pregnancy loss <20 weeks of gestation); stillbirth (intrauterine fetal death ≥20 weeks of gestation). Infant Mortality including; neonatal death (death of a live born infant in the first 28 days of life); infant death (death of an infant after the first 28 days of life). Major congenital anomalies.
Economic Evaluation | From the date of randomization until the infant is 24 months of age (up to 144 weeks)
  A within-trial cost-effectiveness analysis will be conducted comparing costs and outcomes of the trial arms. The analysis will take into account a range of cost items including cost of interventions (i.e., dietary supplements) and cost of eligibility screening. Medicare data and data held by the State departments of health will be used to estimate direct health care costs associated with the management of poor developmental health outcomes over the study period including pharmaceuticals, out of hospital services (e.g., doctor visits), and hospital services (including emergency department presentations).
Urinary Iodine Concentration | At baseline (enrolment <13 weeks of gestation) and mid-pregnancy (28 weeks of gestation)
  At baseline, median iodine concentration by state will be determined to confirm state differences in iodine status that have been previously identified and to determine balance between the two treatment groups. At 28 weeks we will examine median UIC by treatment group to assess group compliance and the success of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Karen P Best, PhD, Principal Investigator — South Australian Health and Medical Research Institute
Locations (1):
- South Australian Health and Medical Research Institute, North Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Yes
Access to study data may be granted, upon review and approval of the HREC, trial steering committee and in accordance with SAHMRI W&K 'Guidelines and Agreement for the use of materials in an ancillary study associated with original clinical trials or cohort studies.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Following final data analysis and primary publication
Access Criteria: Access to study data may be granted, upon review and approval of the HREC, trial steering committee and in accordance with SAHMRI W&K 'Guidelines and Agreement for the use of materials in an ancillary study associated with original clinical trials or cohort studies.

REFERENCES:
- [Derived] Sullivan TR, Green TJ, Gould JF, Makrides MM, Best KP. Statistical analysis plan for the Prenatal Iodine Supplementation and Early Childhood Neurodevelopment (PoppiE) randomised controlled trial. Trials. 2025 May 19;26(1):162. doi: 10.1186/s13063-025-08863-1. PMID 40390018
- [Derived] Best KP, Gould JF, Makrides M, Sullivan T, Cheong J, Zhou SJ, Kane S, Safa H, Sparks A, Doyle LW, McPhee AJ, Nippita TAC, Afzali HHA, Grivell R, Mackerras D, Knight E, Wood S, Green T. Prenatal iodine supplementation and early childhood neurodevelopment: the PoppiE trial - study protocol for a multicentre randomised controlled trial. BMJ Open. 2023 May 10;13(5):e071359. doi: 10.1136/bmjopen-2022-071359. PMID 37164467